CLINICAL TRIAL: NCT01217788
Title: Double Blind Placebo Controlled Study of PH94B for Management of the Symptoms of Generalized Social Phobia
Brief Title: Intranasal PH94B for Management of the Symptoms of Generalized Social Phobia
Acronym: PH94B-SAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pherin Pharmaceuticals, Inc. (Industry)
Responsible Party: Michael R. Liebowitz MD, The Medical Research Network LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH94B CL022
Record Dates: First submitted 2010-09-30; First posted 2010-10-08 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Social Phobia; Social Anxiety Disorder
Keywords: Generalized Social Phobia; Social Anxiety Disorder; Social Phobia; Phobic Disorders; Phobias
MeSH Terms: conditions — Phobia, Social; Phobic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PH94B intranasal spray (Experimental)
  Interventions: Drug: PH94B intranasal spray
- Placebo intranasal spray (Placebo Comparator)
  Interventions: Drug: PH94B intranasal spray

INTERVENTIONS:
Drug: PH94B intranasal spray — Comparison of PH94B single dose intranasal spray and Placebo single dose intranasal spray

SUMMARY:
The purpose of this study is to determine the efficacy of PH94B, a new class of therapeutic compound, administered intranasally for the management of acute anxiety in patients diagnosed with generalized social phobia.

DETAILED DESCRIPTION:
The essential features of generalized social phobia are defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), criteria as a marked and persistent fear of most (generally accepted as four or more) social or performance situations in which the patient believes embarrassment could occur as a consequence of exposure to unfamiliar people and/or possible scrutiny by others. The anxiety resulting from the social or performance situation is profound. The avoidance, fear, or anxious anticipation of these situations interferes significantly with the person's daily routine, having a marked impact on occupational functioning and/or social life. The disorder has a lifetime prevalence estimated at up to 13%, with onset typically in the mid-teens, and it is diagnosed slightly more frequently in females than in males. Social phobia tends to be a chronic disorder with periods of exacerbation, with a reported mean duration of illness of approximately 20 years.

There are two subtypes of social phobia: (i) generalized (discrete), which is suffered by approximately 50% of social phobia patients and in which fear and avoidance extend to a wide range of social situations, and (ii) non-generalized, in which the patient fears only one or a few circumscribed situations. Speaking in front of large groups is by far the most prevalent of social fears (Lang and Stein, 2001).

Social phobia has a lifetime comorbidity rate of approximately 81% with other psychiatric disorders (particularly affective disorders, other anxiety disorders, and substance abuse disorders), as well as to being associated with increased nonpsychiatric medical difficulties. People with social phobia identify social impairment, inadequate social support, overall role impairment, specific impairment in education, work, and other activities, as well as interference in their efforts at self-improvement. Unfortunately, for these patients, there is a strong consensus that social phobia is one of the least commonly recognized and treated mental disorders

ELIGIBILITY:
Inclusion Criteria:

* Subject currently meets the Diagnosis of Social Phobia as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition which is not secondary to another pre-existing psychiatric condition or to a medical condition.
* Liebowitz Social Anxiety Scale (LSAS) score greater than or equal to 60 at Screening.
* Score of 75 or greater on the SUD scale at one of the Performance Phase time points during either the Public Speaking or Social Interaction Challenge
* Written Informed Consent prior to commencing any study specific procedures.
* Women of child-bearing-potential must be able to commit to the consistent and correct use of an acceptable method of birth control throughout the study and have a negative serum pregnancy test result prior to study drug administration.

Exclusion Criteria:

* Use of any psychotropic medication within 30 days prior to study entry.
* Acute or chronic psychiatric disease which is the primary diagnosis (except Social Phobia) at the time of the study. Note that subjects with concurrent Generalized Anxiety Disorder (GAD) are allowed into the study provided this is not the primary diagnosis.
* Subjects with a history of psychiatric diseases such as schizophrenia, bipolar disorder, and psychosis are to be excluded.
* Presence of a clinical condition or disease, or use of a concomitant medication, that in the clinical judgment of the Investigator could place the patient at undue risk, interfere with study participation, or confound the results of the study.
* Use of substances of abuse within the year prior to study entry.
* Concomitant use of any over-the-counter, prescription product, or herbal preparation for treatment of the symptoms of social anxiety during the study and within 30 days prior to study entry and use of non-study anxiolytics such as benzodiazepines during the study and within 30 days prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Subjective Unit of Discomfort Scale | Once before and again 10 minutes after intranasal dosing with PH94B spray, during exposure to a public speaking challenge

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability on the psychometric scale | Once at the end of the intervention and again one week after intervention (follow-up)
  One time after dosing and up to one week after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Liebowitz, M.D., Principal Investigator — Medical Research Network
Locations (1):
- Medical Research Network, New York, New York, United States

REFERENCES:
- [Derived] Liebowitz MR, Salman E, Nicolini H, Rosenthal N, Hanover R, Monti L. Effect of an acute intranasal aerosol dose of PH94B on social and performance anxiety in women with social anxiety disorder. Am J Psychiatry. 2014 Jun;171(6):675-82. doi: 10.1176/appi.ajp.2014.12101342. PMID 24700254